CLINICAL TRIAL: NCT02888015
Title: Does the Use of an Upper Extremity Exercise Program Improve Activity Tolerance and Increase Independence With ADL's
Brief Title: Benefits of Upper Extremity Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 889143-1
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Upper extremity exercise (Other): Five upper extremity exercises will be provided to each of the 10 participants to complete on a daily basis. Exercises included shoulder flexion, elbow flexion/extension, shoulder abduction, internal/external rotation
  Interventions: Other: upper extremity exercise program

INTERVENTIONS:
Other: upper extremity exercise program — five exercises to improve upper extremity strength and endurance will be provided to patients, shoulder flexion, abduction/adduction, elbow flexion/extension, internal/external rotation
  Other Names: exercise program

SUMMARY:
Pt will be provided with a upper extremity exercise program that will be completed daily during their session with occupational therapy. During the session the Activity Measure-Post Acute Care and an activity tolerance chart will be completed. The data from the outcome measures will be used to determine if there is a benefit to completing a daily exercise program.

DETAILED DESCRIPTION:
Study Design This is an evidence-based project based on current research from a literature search. It is a case series design. Patients will be selected from the medical intensive care unit and will be provided with a daily upper extremity exercise program that will be completed in addition to standard interventions such as completion of activities of daily living. Currently therapist within the intensive care unit have the ability to provide upper extremity exercise programs but there is no set standard of care in place for this exercises to be done on a daily basis with patients.

Subject Selection Patients for this project will be selected from the medical intensive care unit at Upstate University Hospital. The physical therapist working in the medical intensive care unit will provide patients with a handout highlighting the project. Patients will be instructed to have their nurse contact the co-investigator through Vocera. Patients will be required to sign a consent form to voluntarily participate in this project. Patients will be expected to engage in an initial evaluation that can take up to an hour. Participation in daily treatment session will also be expected during a patients stay in the hospital. Treatment session can last from 30-60 minutes each day and will continue throughout a patients stay in the medical intensive care unit or a maximum of six weeks, which is the duration of the implementation phase of this project.

Statistical Methods, Data Analysis and Interpretation Quantitative data will be collected through the use of the Activity Measures Post Acute Care, manual muscle testing and the activity-tracking sheet. Information collected from the Activity Measures Post Acute Care will be used to determine if there were improvements in the level of assist for activities of daily living (dressing, bathing, toileting). The scores from the manual muscle testing will be used to determine improvements in upper extremity strength, while the data collected from the activity-tracking chart will be used to see the improvements in activity tolerance. Comparison of data for the manual muscle testing will use information from the initial evaluation and at the time of discharge from the medical intensive care unit. The Activity Measures Post Acute Care and the activity-tracking chart will be performed at each session and data will be compared over the span of the patients stay in the medical intensive care unit.

Study Procedures Pre-Intervention Procedures

* Request and obtain permission from the Director of therapy at Upstate Hospital. Received on 5/31/2016
* Request and obtained permission for the use of the Activity Measure Post Acute Care assessment.
* Completed the CITI training that is a requirement for IRB approval at Upstate Hospital.
* Discuss purpose of the project and review the recruitment handout with Physical therapist in the medical intensive care unit.
* Develop and photocopy recruitment handout for Physical therapist.
* Develop a set of 5 upper extremity exercises that patients will participate in daily developed in Physio-Tools. These exercises will be specialized to clients' needs.

Implementation of project

* The physical therapist on the medical intensive care unit will conduct a physical therapy initial evaluation at which time the patient will be informed of the evidence based project-taking place via a handout provided by the physical therapist.
* The co- investigator will be notified of patient's interest in the project by nursing calling the primary investigator on Vocera.
* The consent interview will be conducted by the co-investigator only. Prior to completion of the initial occupational therapy evaluation, a discussion of the project with the patient will take place to answer any questions that may have come up. Following that discussion participants will sign the informed consent
* The co- investigator will perform an initial occupational therapy evaluation that will assess a patient's ability to complete functional transfers, upper body strength through manual muscle testing and abilities in performing activities of daily living to determine a functional baseline. The outcome measure that will be used to assess activities of daily living is the Activity Measure-Post Acute Care assessment.
* Patients will be provided with an upper extremity exercise program developed in Physio-Tools. Physio Tools has an extensive library of exercises. Each exercise can be customized by number of sets and reps, and by resistance. There will be a set of 5 exercises focused on increasing upper body strength. The 5 exercises chosen will be based off the needs of the patient determined by their scores from the manual muscle testing.
* Patients will be asked to engage in the exercise program on a daily basis during their stay in the intensive care unit. Patients will complete exercises under supervision from the co- investigator during regularly scheduled therapy sessions. During that time patients will be provided with education on proper technique for performing exercises as well as having vitals monitored to ensure safety.
* While completing the exercise program the co- investigator will track the active minutes while the patient is engaged in the exercise and track the inactive minutes while at rest. This will allow for a comparison from session to session to rate if activity tolerance is improving.
* Participants will complete this program one time a day during regular therapy sessions. As their tolerance improves patients may be asked to increase the repetitions and/or may be provided with a resistance band to make it more challenging.
* To complete the whole exercise program should take 30 minutes a session; this time also includes rest breaks. Therapy sessions will take place 5 times a week for the full time that the patient is in the medical intensive care unit.
* The exercise program will be completed each session with the co- investigator. During a therapy session, participants will be asked to engage in activities of daily living. These tasks include dressing, bathing, toileting and grooming.
* During the initial evaluation the patient will determine which activities of daily living they will need to complete in order to be able to safely discharge home. Adaptive equipment for activities of daily living will be provided as needed. To be successful with activities of daily living within the hospital setting, adaptive equipment such as bedside commodes, raised toilet seats and rolling walkers will be provided to assist in achieving independence.
* During this 6 week long project the Activity Measure-Post Acute Care measure, manual muscle testing and the tracking or active and inactive minutest will be completed at each session.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient status on the medical intensive care unit
* Current orders for occupational therapy
* Requires moderate assist or more with 2 or more ADL's based on scores received from the Activity measures post acute assessment tool
* Can follow multiple step commands and are alert and oriented
* Fluent in English
* Individuals 18 years of age and older.

Exclusion Criteria:

* Individuals who are mechanically intubated
* Individuals who the medical team do not feel are medically stable for therapy services
* Individuals receiving continuous veno-venous hemofiltration.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
AM PAC six clicks | 6 weeks
  Addresses six areas of ADL's and information can be gathered by patient report , demonstration of skill or through therapeutic judgment.
Activity tolerance Chart | 6 weeks
  tracking active and inactive minutes during exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Lori Holmes, DPT, Principal Investigator — State University of New York - Upstate Medical University

IPD SHARING:
Plan to Share IPD: No